CLINICAL TRIAL: NCT05345210
Title: Efficacy and Safety of Helicobacter Pylori Eradication Dual or Triple Regimes Using Vonoprazan as the Antacid
Brief Title: Vonoprazan Hp Dual or Triple Eradication Regimes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJLL-KY20222010
Record Dates: First submitted 2022-04-06; First posted 2022-04-25 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Helicobacter Pylori

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Vonoprazan Fumarate+Amoxycillin+Clarithromycin 14days (VAC14) (Active Comparator): Vonoprazan Fumarate 20mg bid po Amoxycillin 1000mg bid po Clarithromycin 500mg bid po for 14 days
  Interventions: Drug: Vonoprazan Fumarate+Amoxycillin+Clarithromycin 14days (VAC14)
- Vonoprazan Fumarate+Amoxycillin 14days (VA14) (Experimental): Vonoprazan Fumarate 20mg bid po Amoxycillin 1000mg bid po for 14 days
  Interventions: Drug: Vonoprazan Fumarate+Amoxycillin 14days (VA14)
- Vonoprazan Fumarate+Amoxycillin 7days (VA7) (Experimental): Vonoprazan Fumarate 20mg bid po Amoxycillin 1000mg bid po for 7 days
  Interventions: Drug: Vonoprazan Fumarate+Amoxycillin 7days (VA7)
- Vonoprazan Fumarate+Tetracycline+Furazolidone 14days (VTF14) (Experimental): Vonoprazan Fumarate 20mg bid po Tetracycline 500mg tid po Furazolidone 100 bid po for 14 days
  Interventions: Drug: Vonoprazan Fumarate+Tetracycline+Furazolidone 14days (VTF14)
- Vonoprazan Fumarate+Tetracycline+Furazolidone 7days (VTF7) (Experimental): Vonoprazan Fumarate 20mg bid po Tetracycline 500mg tid po Furazolidone 100 bid po for 7 days
  Interventions: Drug: Vonoprazan Fumarate+Tetracycline+Furazolidone 7days (VTF7)

INTERVENTIONS:
Drug: Vonoprazan Fumarate+Amoxycillin+Clarithromycin 14days (VAC14) — VAC-14d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po, Clarithromycin 500mg bid po for 14 days VA-14d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po for 14 days VA-7d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po for 7 days VTF-14d:Vonoprazan Fumarate 20mg bid po, Tetracycline 500mg tid po, Furazolidone 100 bid po for 14 days VTF-7d:Vonoprazan Fumarate 20mg bid po, Tetracycline 500mg tid po, Furazolidone 100 bid po for 7 days
  Arms: Vonoprazan Fumarate+Amoxycillin+Clarithromycin 14days (VAC14)
Drug: Vonoprazan Fumarate+Amoxycillin 14days (VA14) — VAC-14d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po, Clarithromycin 500mg bid po for 14 days VA-14d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po for 14 days VA-7d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po for 7 days VTF-14d:Vonoprazan Fumarate 20mg bid po, Tetracycline 500mg tid po, Furazolidone 100 bid po for 14 days VTF-7d:Vonoprazan Fumarate 20mg bid po, Tetracycline 500mg tid po, Furazolidone 100 bid po for 7 days
  Arms: Vonoprazan Fumarate+Amoxycillin 14days (VA14)
Drug: Vonoprazan Fumarate+Amoxycillin 7days (VA7) — VAC-14d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po, Clarithromycin 500mg bid po for 14 days VA-14d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po for 14 days VA-7d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po for 7 days VTF-14d:Vonoprazan Fumarate 20mg bid po, Tetracycline 500mg tid po, Furazolidone 100 bid po for 14 days VTF-7d:Vonoprazan Fumarate 20mg bid po, Tetracycline 500mg tid po, Furazolidone 100 bid po for 7 days
  Arms: Vonoprazan Fumarate+Amoxycillin 7days (VA7)
Drug: Vonoprazan Fumarate+Tetracycline+Furazolidone 14days (VTF14) — VAC-14d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po, Clarithromycin 500mg bid po for 14 days VA-14d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po for 14 days VA-7d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po for 7 days VTF-14d:Vonoprazan Fumarate 20mg bid po, Tetracycline 500mg tid po, Furazolidone 100 bid po for 14 days VTF-7d:Vonoprazan Fumarate 20mg bid po, Tetracycline 500mg tid po, Furazolidone 100 bid po for 7 days
  Arms: Vonoprazan Fumarate+Tetracycline+Furazolidone 14days (VTF14)
Drug: Vonoprazan Fumarate+Tetracycline+Furazolidone 7days (VTF7) — VAC-14d:Vonoprazan Fumarate 20mg bid po, Amoxycillin 1000mg bid po, Clarithromycin 500mg bid po for 14 days
  Arms: Vonoprazan Fumarate+Tetracycline+Furazolidone 7days (VTF7)

SUMMARY:
To evaluate the efficacy and safety of dual or triple regimes for Helicobacter Pylori eradication using Vonoprazan as the antiacid agent.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years old, both gender is eligiable;
* Patients with definite Helicobacter Pylori infection (13C/14C urea breath test, rapid urease test and fecal Helicobacter Pylori antigen test positive) ;
* Voluntary to accept Helicobacter Pylori eradication treatment;
* Females of childbearing age are required to use medically acceptable contraceptive methods during the trial and within 30 days after the trial.

Exclusion Criteria:

* Patients with contraindications to the study drug or allergic to the study drug;
* Severe organ damage and complications (such as liver cirrhosis, uremia, etc.), severe or unstable cardiopulmonary or endocrine diseases;
* Continuous use of anti-ulcer drugs, antibiotics or bismuth complexes (at least 2 weeks before the examination for Helicobacter Pylori infection);
* Pregnant and lactating women;
* Have received upper gastrointestinal surgery;
* Symptoms of dysphagia;
* Evidence of bleeding or iron deficiency anemia;
* have a history of malignant tumor;
* History of drug or alcohol abuse within the past 1 year;
* Systemic application of glucocorticoids, non-steroidal anti-inflammatory drugs, anticoagulants, and platelet aggregation inhibitors (except aspirin ≤100 mg/d);
* Persons with mental disorders;
* Received other clinical trials within the past 3 months;
* Refused to sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter Pylori eradication rate | 28 days after treatment
  The primary end point of this study is H.pylori eradication,established by negative [13C] urea breath test 28 days after the end of eradication

SECONDARY OUTCOMES:
symptoms effective rates | 14 days of treatment, and 28 days after treatment
  symptoms effective rates Evaluation effective rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment. Symptom effective rate =#total score before treatment - total score after treatment#/total score before treatment x100%. Total score = frequency + severity.Frequency score is calculated by all the frequency of heartburn, reflux, abdominal pain, and flatulence. Severity is accumulated by the degree of symptoms described above, which is divided to 4 degree as 0 presenting none, and 3presenting most severe
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache, dizziness, skin rash, other gastrointestinal disorders, pyrexia, cough and back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, Principal Investigator — Xijing Hosipital of Digestive Disease
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No